CLINICAL TRIAL: NCT00142792
Title: Electrical Stimulation for Upper Limb Recovery in Stroke
Brief Title: Functional Electrical Stimulation (FES) for Upper Extremity Recovery in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, John Chae, MD, Prof Vice Chair Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD049777 (NIH); R01HD049777 (NIH)
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Stroke, Acute; Stroke; Hemiparesis
Keywords: stroke; recovery of function; functional electrical stimulation (FES)
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (3):
- A. Cyclic stim (Active Comparator): * Preprogrammed cycles of finger and thumb flexor and extensor stimulation (and flexor stimulation if deemed necessary by the PI) repeatedly and automatically close and open the hand without any effort or voluntary intent required by the subject.
  * Subject instructed to relax, not attempt to assist the stimulation, and not to move the contralateral arm/hand during stimulation
  * Uses NMES device with EMG-triggered and Cyclic capabilities
  Interventions: Device: NMES device with EMG-triggered and Cyclic capabilities
- B. Sensory stim (Active Comparator): Sensory-only electrical stimulation. The stimulation will be cyclic in nature but intensity will be set to a level that can be felt by the patient but not sufficient to cause muscle contraction.
  Uses NMES device with EMG-triggered and Cyclic capabilities
  Interventions: Device: NMES device with EMG-triggered and Cyclic capabilities
- C. EMG-Triggered (Active Comparator): EMG-Triggered electrical stimulation. Subjects in this group will attempt to extend their affected wrist and fingers in response to an audio cue. They will be "rewarded" with stimulation to cause full hand opening once they have generated EMG sufficient to reach a preset threshold level.
  Uses NMES device with EMG-triggered and Cyclic capabilities
  Interventions: Device: NMES device with EMG-triggered and Cyclic capabilities

INTERVENTIONS:
Device: NMES device with EMG-triggered and Cyclic capabilities — All groups will use the NeuroMove NM900 stimulator. Subjects will use the stimulator as described for their group (treatment arm) for two 40-minute sessions per day, 5 days per week for 8 weeks. Surface electrodes for all three groups will be placed over the affected EDC and ECR (finger and wrist extensor) muscles.
  Other Names: NeuroMove NM900 stimulator

SUMMARY:
Stroke is the leading cause of activity limitation among older adults in the United States. NeuroMuscular Electrical Stimulation (NMES) can assist stroke survivors in regaining motor ability and decreasing activity limitation caused by stroke. This study will research the effects of two types of NMES on reducing motor impairment and activity limitation.

DETAILED DESCRIPTION:
Stroke is the leading cause of activity limitation among older adults in the United States. NeuroMuscular Electrical Stimulation (NMES) can be used by stroke survivors who do not have enough residual movement to take part in volitional active repetitive movement therapy and does not require expensive equipment or skilled personnel. Two types of NMES are available. The first is cyclic NMES, which electrically activates paretic muscles at a set duty cycle for a preset time period. (This study will employ both "traditional" cyclic stimulation and "sensory-only" stimulation, in which intensity is set at a level to be felt by the patient but insufficient to cause muscle contraction.)In cyclic NMES, the patient is a passive participant and does not assist the NMES by volitionally contracting the muscle during stimulation. The second type encompasses various forms of NMES in combination with biofeedback. For example, in "EMG-triggered" NMES, subjects are "rewarded" with stimulation in response to successful attempts to reach a pre-set level of EMG activity in the affected muscle. There is increased cognitive input and involvement on the part of the patient. The purpose of this study is to first demonstrate the effectiveness of these two types of surface stimulation on decreasing motor impairment and activity limitation; the study also seeks to assess the effect of adding cognitive input to NMES to reduce motor impairment and activity limitation.

Study subjects will be acute stroke survivors. They will participate for a total of eight months, beginning within the first six months after their stroke. Subjects will be randomly assigned to one of three treatment groups and will receive stimulation accordingly: 1) Cyclic stimulation; 2)Sensory-only stimulation; and 3)EMG-triggered stimulation. Members of each treatment group will be given an appropriate NMES device to use for two 40-minute treatment sessions per day, five times per week for eight weeks; for a total of 80 treatment sessions. Stimulation will be applied to ECR and EDC (wrist and finger extensors) on the affected arm. A treatment therapist will visit the patient at home on a weekly basis to monitor subject compliance and to provide feedback on device usage. The primary outcome measure will be the upper extremity portion of the Fugl-Meyer Motor Assessment (FMA), a measure of motor impairment. The modified Arm Motor Ability Test (mAMAT) is a hemiparetic arm-specific measure of activity limitation, and will serve as a secondary outcome measure.

In addition to the baseline visit on day of enrollment, subjects will complete these outcome measurements at the clinic on five other occasions: at mid-treatment (week 5); end of treatment (week 9); and for follow-up visits at one-, three- and six-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-89
* Evidence of clinical symptoms from a hemorrhagic or nonhemorrhagic stroke with all symptoms from previous stroke(s) completely resolved
* Medically stable
* Less than 6 months post-stroke
* Intact skin on the hemiparetic side
* Able to follow 3-stage commands
* Able to recall 2/3 objects after 30 minutes
* Full passive ROM at the wrist and the thumb, index and long finger MCP joints on the affected side
* Presence of a detectable, volitionally-activated EMG signal from the paretic wrist or finger extensors (ECR or EDC)
* Affected wrist extensors ≤ 4 on MRC scale
* Score of ≤ 11/14 on Section C (hand) of UE portion of Fugl Meyer Assessment (FMA)
* Ability to tolerate NMES to the ECR and EDC for full wrist and finger extension
* Caregiver available to assist with the device every day (unless subject capable of using it independently

Exclusion Criteria:

* History of ventricular arrythmias or any other arrythmias (i.e. fast atrial fibrillation, ventricular tachycardia, or supraventricular tachycardia) with hemodynamic instability
* History of other upper motor neuron lesion
* Absent sensation of the affected limb
* Pregnancy
* History of more than one seizure per month during the last year (or, since the stroke if no seizures prior to stroke)
* Discharge to a skilled nursing facility or long-term care facility (EXCEPTION: Subjects may be d/c'd to the 6A SNF unit at MetroHealth Medical Center)
* Uncompensated hemineglect
* Implanted stimulator (such as a pacemaker)
* Evidence of hand pain as defined by current metacarpophalangeal (MCP) joint pain upon palpation and/or wrist or MCP pain upon extension

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2005-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Chae, MD, Principal Investigator — MetroHealth Medical Center
Locations (3):
- United States (3):
  - Edwin Shaw Rehab - Akron General Medical Center, Akron, Ohio
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glanz M, Klawansky S, Stason W, Berkey C, Chalmers TC. Functional electrostimulation in poststroke rehabilitation: a meta-analysis of the randomized controlled trials. Arch Phys Med Rehabil. 1996 Jun;77(6):549-53. doi: 10.1016/s0003-9993(96)90293-2. PMID 8831470
- [Background] Chae J, Bethoux F, Bohine T, Dobos L, Davis T, Friedl A. Neuromuscular stimulation for upper extremity motor and functional recovery in acute hemiplegia. Stroke. 1998 May;29(5):975-9. doi: 10.1161/01.str.29.5.975. PMID 9596245
- [Background] Powell J, Pandyan AD, Granat M, Cameron M, Stott DJ. Electrical stimulation of wrist extensors in poststroke hemiplegia. Stroke. 1999 Jul;30(7):1384-9. doi: 10.1161/01.str.30.7.1384. PMID 10390311
- [Background] Francisco G, Chae J, Chawla H, Kirshblum S, Zorowitz R, Lewis G, Pang S. Electromyogram-triggered neuromuscular stimulation for improving the arm function of acute stroke survivors: a randomized pilot study. Arch Phys Med Rehabil. 1998 May;79(5):570-5. doi: 10.1016/s0003-9993(98)90074-0. PMID 9596400
- [Background] Cauraugh J, Light K, Kim S, Thigpen M, Behrman A. Chronic motor dysfunction after stroke: recovering wrist and finger extension by electromyography-triggered neuromuscular stimulation. Stroke. 2000 Jun;31(6):1360-4. doi: 10.1161/01.str.31.6.1360. PMID 10835457
- [Background] Cauraugh JH, Kim S. Two coupled motor recovery protocols are better than one: electromyogram-triggered neuromuscular stimulation and bilateral movements. Stroke. 2002 Jun;33(6):1589-94. doi: 10.1161/01.str.0000016926.77114.a6. PMID 12052996
- [Background] Sonde L, Gip C, Fernaeus SE, Nilsson CG, Viitanen M. Stimulation with low frequency (1.7 Hz) transcutaneous electric nerve stimulation (low-tens) increases motor function of the post-stroke paretic arm. Scand J Rehabil Med. 1998 Jun;30(2):95-9. doi: 10.1080/003655098444192. PMID 9606771
- [Background] Sonde L, Kalimo H, Fernaeus SE, Viitanen M. Low TENS treatment on post-stroke paretic arm: a three-year follow-up. Clin Rehabil. 2000 Feb;14(1):14-9. doi: 10.1191/026921500673534278. PMID 10688340
- [Background] Bowman BR, Baker LL, Waters RL. Positional feedback and electrical stimulation: an automated treatment for the hemiplegic wrist. Arch Phys Med Rehabil. 1979 Nov;60(11):497-502. PMID 508075
- [Background] Kraft GH, Fitts SS, Hammond MC. Techniques to improve function of the arm and hand in chronic hemiplegia. Arch Phys Med Rehabil. 1992 Mar;73(3):220-7. PMID 1543423
- [Background] Kimberley TJ, Lewis SM, Auerbach EJ, Dorsey LL, Lojovich JM, Carey JR. Electrical stimulation driving functional improvements and cortical changes in subjects with stroke. Exp Brain Res. 2004 Feb;154(4):450-60. doi: 10.1007/s00221-003-1695-y. Epub 2003 Nov 15. PMID 14618287
- [Derived] Wilson RD, Page SJ, Delahanty M, Knutson JS, Gunzler DD, Sheffler LR, Chae J. Upper-Limb Recovery After Stroke: A Randomized Controlled Trial Comparing EMG-Triggered, Cyclic, and Sensory Electrical Stimulation. Neurorehabil Neural Repair. 2016 Nov;30(10):978-987. doi: 10.1177/1545968316650278. Epub 2016 May 24. PMID 27225977
- See also: Cleveland FES Center — http://fescenter.org/index.php
- See also: The MetroHealth System - Clinical Trials — http://www.metrohealth.org/body.cfm?id=2438
- See also: Neuromotor Recovery & Rehabilitation Laboratory, Cincinnati, Ohio — http://rehablab.org

RESULTS

PARTICIPANT FLOW:
Groups:
- A. Cyclic Stim: * Preprogrammed cycles of finger and thumb flexor and extensor stimulation (and flexor stimulation if deemed necessary by the PI) repeatedly and automatically close and open the hand without any effort or voluntary intent required by the subject.
  * Subject instructed to relax, not attempt to assist the stimulation, and not to move the contralateral arm/hand during stimulation
  NMES device with EMG-triggered and Cyclic capabilities: All groups will use the NeuroMove NM900 stimulator. Subjects will use the stimulator as described for their group (treatment arm) for two 40-minute sessions per day, 5 days per week for 8 weeks. Surface electrodes for all three groups will be placed over the affected EDC and ECR (finger and wrist extensor) muscles.
- C. EMG-Triggered: EMG-Triggered electrical stimulation. Subjects in this group will attempt to extend their affected wrist and fingers in response to an audio cue. They will be "rewarded" with stimulation to cause full hand opening once they have generated EMG sufficient to reach a preset threshold level.
  NMES device with EMG-triggered and Cyclic capabilities: All groups will use the NeuroMove NM900 stimulator. Subjects will use the stimulator as described for their group (treatment arm) for two 40-minute sessions per day, 5 days per week for 8 weeks. Surface electrodes for all three groups will be placed over the affected EDC and ECR (finger and wrist extensor) muscles.
- B. Sensory Stim: Sensory-only electrical stimulation. The stimulation will be cyclic in nature but intensity will be set to a level that can be felt by the patient but not sufficient to cause muscle contraction.
  NMES device with EMG-triggered and Cyclic capabilities: All groups will use the NeuroMove NM900 stimulator. Subjects will use the stimulator as described for their group (treatment arm) for two 40-minute sessions per day, 5 days per week for 8 weeks. Surface electrodes for all three groups will be placed over the affected EDC and ECR (finger and wrist extensor) muscles.
Period: Overall Study
Arm/Group | A. Cyclic Stim | C. EMG-Triggered | B. Sensory Stim
Started | 39 | 41 | 42
Completed Intervention | 35 | 37 | 37
Completed | 27 | 26 | 30
Not Completed | 12 | 15 | 12
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 3
Not completed — Lost to Follow-up | 8 | 11 | 7
Not completed — No category | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Non-hospitalized adults within 6 months of stroke aged 21-89 years.
Groups:
- Total: Total of all reporting groups
Arm/Group | A. Cyclic Stim | C. EMG-Triggered | B. Sensory Stim | Total
Number analyzed (Participants) | 39 | 41 | 42 | 122
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55.0 [47.4 to 65.9] | 58.6 [48.9 to 67.5] | 55.8 [47.6 to 66.7] | 55.1 [47.6 to 67.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 16 | 51
  Male | 21 | 24 | 26 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 38 | 40 | 41 | 119
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 14 | 9 | 32
  White | 30 | 27 | 30 | 87
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 39 | 41 | 42 | 122
Months from Stroke [Median (Inter-Quartile Range); unit: months] | 2.0 [1.3 to 4.2] | 2.9 [1.5 to 4.7] | 3.2 [1.7 to 5.0] | 2.8 [1.5 to 4.5]

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Motor Assessment (FMA) - Motor Impairment Measure
Description: The FMA battery measures six dimensions of post-stroke impairment including upper and lower limb motor impairment, range of motion, pain, reflexes, and sensation. , "Each item (33 total) is graded on a 3-point ordinal scale (0, cannot perform; 1, perform partially; and 2, perform fully) and summed to provide a score ranging from 0 to 66, where higher scores indicate better motor function The FMA was administered with the participant seated.
Time Frame: FMA will be administered on 6 occasions: at baseline, mid-treatment, end of treatment, and follow-up at 1-,3- and 6-months post-treatment.
Population: All cases, intent-to-treat, adjusted for site
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A. Cyclic Stim | C. EMG-Triggered | B. Sensory Stim
Number analyzed (Participants) | 39 | 41 | 42
units on a scale
  Baseline | 27.5 [23.4 to 31.6] | 29.8 [25.7 to 33.9] | 26.8 [22.9 to 30.6]
  Mid Treatment | 31.8 [27.6 to 36.1] | 32.6 [28.2 to 37.0] | 30.4 [26.4 to 34.4]
  End of Treatment | 34.6 [30.5 to 38.7] | 34.7 [30.0 to 39.5] | 33.6 [29.1 to 38.1]
  1 month after treatment | 33.6 [31.1 to 39.6] | 36.3 [31.7 to 41.0] | 35.2 [30.4 to 39.9]
  3 months after treatment | 37.9 [33.6 to 42.1] | 39.3 [34.4 to 44.2] | 37.3 [32.8 to 41.8]
  6 months after treatment | 39.3 [34.8 to 43.8] | 39.5 [34.7 to 44.3] | 37.6 [32.6 to 42.5]
Statistical Analysis 1: Comparison: A. Cyclic Stim vs C. EMG-Triggered vs B. Sensory Stim; The study was powered to detect differences in FMA scores of a minimum effect size of 0.8 at a significance level of 0.01, the smallest effect size difference anticipated between Cyclic NMES and Cyclic Sensory Stimulation based on prior studies. A significance level of 0.01 in the power-analysis was taken since for each measurement occasion, three post-hoc tests are needed. To account for drop out of 20 % , the minimum number of participants required per group is 63; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis — Time by group interaction effect, F(2,372) = 1.8, p =0.18); A random intercept for each participant with a first-order antedependent covariance structure. Adjusted for site
Statistical Analysis 2: Comparison: A. Cyclic Stim vs C. EMG-Triggered vs B. Sensory Stim; Test type: Superiority; p < 0.001, Mixed Models Analysis — time effect, F(1,109)=87.7, p<0.001); A random intercept for each participant with a first-order antedependent covariance structure. Adjusted for site

2. Secondary Outcome: Arm Motor Ability Test (AMAT) - Hemiparetic Arm-specific Measure of Activity Limitation
Description: The AMAT assesses upper limb specific tasks and does not allow for compensation. The AMAT consists of 13 compound ADL tasks composed of 1 to 3 component tasks, with a total of 28 component tasks. Each task was rated on the functional ability ordinal scale from 0-5 and an average is calculated, so the final score remains 0-5, with higher scores indicating lesser activity limitation. Total range of reported data is between 0 and 5 because the average is reported. 0 refers to no function. 5 refers to normal function.
Time Frame: AMAT will be administered on 6 occasions as above: at baseline, mid-treatment, end of treatment, and follow-up at 1-,3- and 6-months post-treatment.
Population: All cases, intent to treat
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A. Cyclic Stim | C. EMG-Triggered | B. Sensory Stim
Number analyzed (Participants) | 39 | 41 | 42
units on a scale
  Baseline | 1.7 [1.4 to 2.0] | 2.0 [1.6 to 2.4] | 1.7 [1.3 to 2.0]
  Mid Treatment | 2.2 [1.9 to 2.6] | 2.3 [1.9 to 2.7] | 2.0 [1.6 to 2.3]
  End of Treatment | 2.4 [2.0 to 2.8] | 2.4 [2.0 to 2.9] | 2.1 [1.7 to 2.5]
  1 month after treatment | 2.6 [2.2 to 3.0] | 2.5 [2.1 to 3.0] | 2.3 [2.0 to 2.7]
  3 months after treatment | 2.7 [2.3 to 3.1] | 2.8 [2.3 to 3.2] | 2.5 [2.1 to 2.9]
  6 months after treatment | 2.9 [2.5 to 3.4] | 2.8 [2.3 to 3.2] | 2.7 [2.2 to 3.1]
Statistical Analysis 1: Comparison: A. Cyclic Stim vs C. EMG-Triggered vs B. Sensory Stim; Test type: Superiority or Other; p = 0.27, Mixed Models Analysis — time by group interaction effect, F(2,373) = 1.3, p =0.27; A random intercept for each participant with a first-order antedependent covariance structure. Adjusted for site
Statistical Analysis 2: Comparison: A. Cyclic Stim vs C. EMG-Triggered vs B. Sensory Stim; Test type: Superiority; p < 0.001, Mixed Models Analysis — time effect, F(1,109)=91.1, p<0.001; A random intercept for each participant with a first-order antedependent covariance structure. Adjusted for site

ADVERSE EVENTS:
Arm/Group | A. Cyclic Stim | C. EMG-Triggered | B. Sensory Stim
Serious Adverse Events (participants affected / at risk) | 10/39 | 13/41 | 9/42
Other Adverse Events (participants affected / at risk) | 1/39 | 3/41 | 2/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A. Cyclic Stim (N=39) | C. EMG-Triggered (N=41) | B. Sensory Stim (N=42)
Illness, +/- hospitalization (General disorders) | 5 (8) | 7 (7) | 5 (5)
Fall (General disorders) | 2 (2) | 0 (0) | 1 (1)
Surgery or procedure (Investigations) | 1 (1) | 4 (5) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Other (General disorders) | 4 (4) | 6 (7) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A. Cyclic Stim (N=39) | C. EMG-Triggered (N=41) | B. Sensory Stim (N=42)
Shock (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2) — Subjects received non-injurious electrical stimulus while moving electrode pads when stimulator was in operation
Muscle Twitch (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Subject experienced muscle twitching other than expected

LIMITATIONS AND CAVEATS:
the estimated sample size needed to reach 90% power to detect clinically meaningful differences within the groups was not met due to slow recruitment. The lower power creates the possibility that a type II error was made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No